CLINICAL TRIAL: NCT00387036
Title: A Multicenter, Double-Blind Placebo-Controlled Crossover Study to Investigate the Effects of an Inhaled Corticosteroid on Cardiopulmonary Exercise Parameters in Patients With Chronic Obstructive Pulmonary Disease
Brief Title: Exercise Study in Patient With Chronic Obstructive Pulmonary Disease (0000-036)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Termininated for business reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0000-036; 036; 2006_039
Record Dates: First submitted 2006-10-05; First posted 2006-10-12 (Estimated); Results first posted 2010-05-26 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Other): Arm 1: drug, crossing over to Pbo comparator
  Interventions: Drug: Fluticasone
- 2 (Other): Arm 2: Pbo comparator, crossing over to drug
  Interventions: Drug: Fluticasone; Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Fluticasone — fluticasone 250 µg/inhalation, 2 inhalations bid. 14 Days of treatment.
Drug: Comparator: Placebo — Placebo /inhalation, 2 inhalations bid. 14 Days of treatment.
  Arms: 2

SUMMARY:
To test the effect of the research study drug, inhaled fluticasone on lung function in exercising patients with Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* 40 years and older
* Clinical diagnosis of COPD for greater than one year
* History of cigarette smoking

Exclusion Criteria:

* Other lung diseases (not including COPD), such as asthma
* A condition that could interfere with your ability to perform exercise tests

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-12; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Result] Guenette JA, Raghavan N, Harris-McAllister V, Preston ME, Webb KA, O'Donnell DE. Effect of adjunct fluticasone propionate on airway physiology during rest and exercise in COPD. Respir Med. 2011 Dec;105(12):1836-45. doi: 10.1016/j.rmed.2011.08.021. Epub 2011 Sep 13. PMID 21917440

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 1 center in Canada.
  Patient screening began 14-Dec-2006 and the first patient was randomized on 16-Feb-2007.
  Last patient last visit for the study was 31-Jul-2009.
Pre-assignment Details: Patients must have met the following criteria: FEV1 (Forced expiratory volume in 1 second) less than or equal to (≤) 70% and FEV1/ FVC (forced vital capacity) ≤ to 0.7; FRC (functional residual capacity) greater than or equal to (≥)120% of the predicted value, and moderate to severe chronic activity-related dyspnea ≥ 120% of the predicted value.
Groups:
- Fluticasone Propionate Then Placebo: Following 1 week Placebo run-in period (Period I), patients were randomized to receive fluticasone propionate 250 mcg Hydrofluoroalkane (HFA) 2 inhalations twice daily for a 2-week period (Period II) followed by 2-week washout period (Period III) and 2-week placebo 2 inhalations twice daily (Period IV).
- Placebo Then Fluticasone Propionate: Following 1 week Placebo run-in period (Period I), patients were randomized to receive placebo 2 inhalations twice daily for a 2-week period (Period II) followed by 2-week washout period (Period III) and 2-week fluticasone propionate 250 mcg HFA 2 inhalations twice daily (Period IV).
Period: 2-Week First Intervention
Arm/Group | Fluticasone Propionate Then Placebo | Placebo Then Fluticasone Propionate
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: 2-Week Placebo Washout
Arm/Group | Fluticasone Propionate Then Placebo | Placebo Then Fluticasone Propionate
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: 2-Week Crossover Second Intervention
Arm/Group | Fluticasone Propionate Then Placebo | Placebo Then Fluticasone Propionate
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Arm/Group | Entire Study Population
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 8
Exercise endurance time at the beginning of Fluticasone Propionate [Mean (Standard Deviation); unit: Minutes] — The duration of loaded pedaling at the beginning of Fluticasone Propionate treatment.
  Minutes | 9.67 (7.88)
Exercise endurance time at the beginning of placebo treatment [Mean (Standard Deviation); unit: Minutes] — The duration of loaded pedaling at the beginning of placebo treatment
  Minutes | 9.42 (6.73)
Standardized Dyspnea Score at isotime at the beginning of Fluticasone [Mean (Standard Deviation); unit: Units on a Scale] — Standardized Dyspnea Score (0 (no discomfort) to 10 (most severe)) at isotime at the beginning of Fluticasone Propionate treatment. Isotime is the duration of the shortest exercise test on all treatment days (or the longest exercise time point common to all constant-load exercise tests).
  Units on a Scale | 4.50 (1.87)
Standardized Dyspnea Score at isotime at the beginning of placebo [Mean (Standard Deviation); unit: Units on a Scale] — Standardized Dyspnea Score (0 (no discomfort) to 10 (most severe)) at isotime at the beginning of placebo treatment. Isotime is the duration of the shortest exercise test on all treatment days (or the longest exercise time point common to all constant-load exercise tests)
  Units on a Scale | 4.75 (2.13)

OUTCOME MEASURES:

1. Primary Outcome: Standardized Dyspnea Score at Isotime During Exercise
Description: Difference in standardized dyspnea rating at isotime during constant load exercise in patients with COPD between Fluticasone Propionate treatment and placebo treatment at the end of the treatment period.
  Isotime is the duration of the shortest exercise test on all treatment days (or the longest exercise time point common to all constant-load exercise tests). The standardized dyspnea score will be measured with the modified 10-point Borg Scale (0 [Best] - 10 [Worst] ).
Time Frame: 2 Weeks
Population: Intention to treat analysis. All patients were included.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Groups:
- Fluticasone Propionate: Fluticasone Propionate 250 mcg HFA (hydrofluoroalkane) administered 2 inhalations twice daily in first or second intervention
- Placebo: Placebo administered 2 inhalations twice daily in first or second intervention
Arm/Group | Fluticasone Propionate | Placebo
Number analyzed (Participants) | 12 | 12
Units on a Scale | 3.58 (2.14) | 4.50 (2.18)
Statistical Analysis 1: Comparison: Fluticasone Propionate vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = -0.92, 90% CI [-1.59 to -0.25], Standard Error of Mean 0.37

2. Secondary Outcome: Exercise Endurance Time
Description: Difference in exercise endurance time between Fluticasone Propionate treatment and placebo treatment at the end of the treatment period.
Time Frame: 2 Weeks
Population: Intention to treat analysis. All patients were included.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Fluticasone Propionate | Placebo
Number analyzed (Participants) | 12 | 12
Minutes | 12.92 (10.52) | 9.75 (6.93)
Statistical Analysis 1: Comparison: Fluticasone Propionate vs Placebo; Test type: Superiority or Other; Mean Difference (Final Values) = 3.17, 90% CI [-0.28 to 6.61], Standard Error of Mean 1.90

ADVERSE EVENTS:
Time Frame: Screening to 14 days after last dose of study medication.
Arm/Group | Fluticasone Propionate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 5/12 | 2/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fluticasone Propionate (N=12) | Placebo (N=12)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Infection (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
Viral Infection (Infections and infestations) | 1 | 0
Tooth Fracture (Injury, poisoning and procedural complications) | 1 | 0
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper Respiratory Tract Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.